CLINICAL TRIAL: NCT01240278
Title: Pilot Study to Examine Histological Characteristics of Mammographic Density With Molecular Breast Imaging: Part 1 - Postmenopausal Women
Brief Title: Histology of Functional Density in Postmenopausal Breast
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Carrie Hruska, Professor, Mayo Clinic
Other Study IDs: 10-004506
Record Dates: First submitted 2010-11-05; First posted 2010-11-15 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Dense Breasts; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — core biopsy samples of dense breast tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Increased mammographic density is recognized as an important risk factor for developing breast cancer, however, the underlying mechanism explaining this relationship is unclear. The investigators hypothesize that Molecular Breast Imaging (MBI) can more accurately distinguish dense tissue on mammography which is at high risk from dense tissue at low risk by indicating cellular activity in dense tissue as radiotracer uptake (functional density) in the breast. In this pilot study, the investigators want to compare the histological characteristics of breast tissue in patients with who have similar density on mammography but different levels of functional density on MBI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 or older
2. Be postmenopausal as defined as having at least 12 consecutive months of amenorrhea
3. Screening mammogram performed at Mayo Clinic Rochester within one year prior to the current MBI study which demonstrates

   1. Negative or benign assessment (BIRADs category 1-2)
   2. No proliferative benign lesions (e.g. fibroadenomas) identified
   3. Heterogeneously dense or extremely dense parenchyma (BIRADs density category 3 or 4)
4. MBI performed less than one month prior to biopsy demonstrating either significant FD or photopenic FD.

Exclusion criteria:

1. Using any exogenous hormones (e.g., hormonal contraceptives, sex steroid hormones) or any estrogen receptor modulating drugs (e.g., tamoxifen, raloxifene) or any aromatase inhibitors within six months prior to study biopsy.
2. Personal history of any cancer, except non-melanomatous skin cancer
3. Current breast symptoms
4. Breast implants
5. Known allergy to local anesthetic.
6. History of bleeding complications from prior interventions
7. Current use of anticoagulants (e.g., Coumadin or other blood thinners)
8. Major medical condition

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with mammographically dense breasts who demonstrate either photopenic or marked background parenchymal uptake on MBI.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
proportion of epithelium vs stroma | within 1 month of functional density assessment on MBI

SECONDARY OUTCOMES:
Degree of lobular involution | within 1 month of functional density assessment on MBI
  Degree of lobular involution as assessed through qualitative and quantitative measurements will be compared between dense tissue which appears photopenic on MBI and dense tissue which appears functionally active on MBI.
Ki-67 cellular proliferation index | within 1 month of functional density assessment on MBI
  Degree of cellular proliferation as assessed through Ki-67 index will be compared between dense tissue which appears photopenic on MBI and dense tissue which appears functionally active on MBI.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Hruska, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bardwell Speltz L, Ghosh K, Visscher DW, Scott CG, Cole KC, Kroneman TN, Maxwell RW, Conners AL, Hunt KN, Rhodes DJ, Vachon CM, Hruska CB. Histologic correlates of background parenchymal uptake on molecular breast imaging. Breast Cancer Res. 2025 Dec 16;27(1):216. doi: 10.1186/s13058-025-02171-x. PMID 41402965
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials